CLINICAL TRIAL: NCT03375359
Title: First Trimester Screening for Trisomy 21, 18, 13 and 22q11.2 Deletion Syndrome - ReFaPo02
Brief Title: Reducing False Positives in Prenatal Screening
Acronym: ReFaPo02
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: PerFet_ReFaPo02
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
MeSH Terms: interventions — Noninvasive Prenatal Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cfDNA screening: Pregnant women who are referred for FTS or for further follow-up examinations in case of a suspected anomaly or increased nuchal translucency at 11-13 weeks' gestation can be recruited for this study.
  Interventions: Diagnostic Test: cfDNA screening

INTERVENTIONS:
Diagnostic Test: cfDNA screening — cfDNA screening test for aneuploidy risk assessment

SUMMARY:
Combined first-trimester screening represents the gold standard of risk assessment for the presence of trisomy 21, 18, and 13. The concept is based on the age risk, the measurement of fetal nuchal translucency (NT), and the determination of serum markers free beta-hCG and PAPP-A in maternal blood.

In recent years it has been shown that the risk assessment can be improved by combining in-depth ultrasound and cell-free DNA analysis from maternal blood. In their latest study, the investigators were able to detect all fetuses with trisomy 21, 18, and 13 through this procedure. No normal fetus displayed an increased risk. In contrast, the detection rate in classic, combined first-trimester screening is about 95% and the false-positive rate is 3-5%. In this study the investigator examine the test quality - especially the false positives - of cell-free DNA analysis on trisomy 21, 18 and 13 as well as on the microdeletion 22q in 1000 pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age of 18 years and more
* Crown rump length 45 - 84mm
* Referral for first trimester risk assessment
* Singleton pregnancy
* Written consent

Exclusion Criteria:

* No consent
* Known parental microdeletion 22q11.2
* Crown rump length <45mm or >84mm
* Multiple pregnancies including vanishing twins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are referred for FTS or for further follow-up examinations in case of a suspected anomaly or increased nuchal translucency at 11-13 weeks' gestation
Sampling Method: Non-Probability Sample
Enrollment: 1127 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Screen positive rate | 15 month
  Screen-positive rate will be calculated by proportion of high risk results compared to all cfDNA tests performed
Screen false-positive rate | 15 month
  False-positive rate will be calculated by proportion of high risk results compared to all cfDNA tests performed in pregnancies with a normal offspring
Uninformative test rate in cfDNA screening for 22q11.2 deletion | 15 month
  Rate of uninformative tests will be defined by proportion of cfDNA screening for 22q11.2 deletion without results compared to all cfDNA tests performed

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Oliver Kagan, Prof., Principal Investigator — University Hospital Tuebingen, Department of Women's Health
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany